CLINICAL TRIAL: NCT05993195
Title: Comparative Analysis of Re-operation Rates of Concorde Bullet Device Versus Conduit Titanium Interbody Graft for Lumbar Fusion
Brief Title: Re-operation Rates of Concorde Bullet Device Versus Conduit Titanium Interbody Graft for Lumbar Fusion
Status: Completed | Type: Observational
Sponsor: Lahey Clinic (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Sponsor
Other Study IDs: 20213046
Record Dates: First submitted 2023-06-14; First posted 2023-08-15 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Degenerative Spondylolisthesis; Lumbar Spondylosis; Lumbar Spondylolisthesis
Keywords: lumbar fusion
MeSH Terms: conditions — Spondylosis; Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Conduit Interbody device: The Conduit Titanium Interbody Graft will be compared to the Concorde Bullet Device group for PLIF and TLIF.
  Interventions: Device: Conduit Titanium Interbody Graft
- Concorde Bullet Device: The control group is patients with degenerative spondylotic disease undergoing either one level or two level fusions with Concorde Bullet Device interbody device.
  Interventions: Device: Concorde Bullet Device

INTERVENTIONS:
Device: Conduit Titanium Interbody Graft — The Concorde Bullet Device is compared with Conduit Titanium Interbody Graft for lumber fusion in terms of reoperation rates at 2 years.
  Groups: Conduit Interbody device
Device: Concorde Bullet Device — This traditional device is to compare the clinical results of the new Conduit Titanium Interbody device for lumbar fusion
  Groups: Concorde Bullet Device

SUMMARY:
The purpose of this early study is to compare the clinical results of the new Conduit Interbody device to the traditional Concorde Bullet Device. The primary objective is to explore the rates and reasons for re-operation between both constructs at 2 years.

DETAILED DESCRIPTION:
The demand for lumbar fusion continues to rise with the growing and aging population. Additionally, new and innovative technologies continue to bring new devices to the market. However, our understanding of how emerging constructs compare with existing technology is lacking. The purpose of this study is to compare the clinical results of the new Conduit Interbody device to the traditional Concorde Bullet Device in lumbar fusion, one or two levels between L2-S1 will be included. Both transforaminal lumbar interbody fusion (TLIF) and posterior lumbar interbody fusion (PLIF) approaches will be included in the patient cohort. The primary objective is to explore the rates and reasons for re-operation between both constructs at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older with symptomatic degenerative lumbar spondylotic disease, either spondylosis, and/or spondylolisthesis
* who have failed conservative management of at least 6 weeks requiring 1 or 2 level lumbar interbody fusion (either PLIF or TLIF)
* All patients included will be index surgeries (no re-operations).

Exclusion Criteria:

* Patients who improve with consecutive management and do not undergo lumbar fusion surgery
* Surgery performed in the thoracic or cervical spine
* Surgery performed for tumor, infection, or trauma Patients who have an unstable fracture, tumor, and osteoporosis with T score exceeding -2.0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion of interbody devices resulted in higher of lumbar fusion, however, new devices have not been fully evaluated clinical and radiographically in terms of overall outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Reoperation rate | 1 year and at 2 years
  a comparison of Concorde Bullet Device versus Conduit Titanium Interbody Graft for lumbar fusion in terms of reoperation rate

SECONDARY OUTCOMES:
Surgical Variables of Concorde Bullet Device versus Conduit Titanium Interbody Graft for lumber fusion | 2 years
  Assessment of surgical variables, such as type of bone graft or bone graft extenders (including ViviGen, bone morphogenetic protein (BMP), tricalcium phosphate, local autograft, allograft, allograft chips, or demineralized bone matrix), on reoperations

OTHER OUTCOMES:
Baseline Demographics of Concorde Bullet Device versus Conduit Titanium Interbody Graft for lumber fusion | 1 year and 2 years
  Demographics, comorbidities, will be assessed including efficacy, safety, and fusion rates.
  Demographics include the following: gender, age, race, BMI, weight (oz.), height (inches), ASA class, surgery level.
  Comorbidities include the following: diabetes, heart failure, coronary artery disease, anxiety/depression, active smoker, pre-operative opioid use.
EQ5D of Concorde Bullet Device versus Conduit Titanium Interbody Graft for lumber fusion | 1 year and 2 years
  The EQ5D index scale is a 5-dimension standardized measurement of heath status developed by EuroQol. The EQ5D index is derived by applying a formula that consist of weights. It is calculated by assigning a numerical value to each response level (ie. 1 for "no problem", 3 for "extreme problem"/"unable to"). The EQ5D scale ranges from 0 (worst imaginable health state) to 100 (best imaginable health scale).
ODI of Concorde Bullet Device versus Conduit Titanium Interbody Graft for lumber fusion | 1 year and 2 years
  The Oswestry Disability Index is a gold standard outcome measure that was designed to assess daily function for those who experience back pain. The questionnaire consists of 10 questions presented as a 6-Likert scale. For each section the total possible score is 5; the first statement marked would score=0; the last statement marked would score=5. Scores range from 0% to 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Whitmore, MD, FAANS, Principal Investigator — Lahey Hospital & Medical Center; Edilin Lopez, MD, Study Director — Lahey Hospital & Medical Center
Locations (1):
- Lahey Hospital and Medical Center, Burlington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with DePuy Synthes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 years
Access Criteria: The data is accessed only by the study sponsor.

REFERENCES:
- [Background] Greiner-Perth R, Boehm H, Allam Y, Elsaghir H, Franke J. Reoperation rate after instrumented posterior lumbar interbody fusion: a report on 1680 cases. Spine (Phila Pa 1976). 2004 Nov 15;29(22):2516-20. doi: 10.1097/01.brs.0000144833.63581.c1. PMID 15543064
- [Background] Irmola TM, Hakkinen A, Jarvenpaa S, Marttinen I, Vihtonen K, Neva M. Reoperation Rates Following Instrumented Lumbar Spine Fusion. Spine (Phila Pa 1976). 2018 Feb 15;43(4):295-301. doi: 10.1097/BRS.0000000000002291. PMID 28614279
- [Background] Choudhri TF, Mummaneni PV, Dhall SS, Eck JC, Groff MW, Ghogawala Z, Watters WC 3rd, Dailey AT, Resnick DK, Sharan A, Wang JC, Kaiser MG. Guideline update for the performance of fusion procedures for degenerative disease of the lumbar spine. Part 4: radiographic assessment of fusion status. J Neurosurg Spine. 2014 Jul;21(1):23-30. doi: 10.3171/2014.4.SPINE14267. PMID 24980581
- [Background] Carreon LY, Djurasovic M, Glassman SD, Sailer P. Diagnostic accuracy and reliability of fine-cut CT scans with reconstructions to determine the status of an instrumented posterolateral fusion with surgical exploration as reference standard. Spine (Phila Pa 1976). 2007 Apr 15;32(8):892-5. doi: 10.1097/01.brs.0000259808.47104.dd. PMID 17426635
- [Background] Carreon LY, Glassman SD, Schwender JD, Subach BR, Gornet MF, Ohno S. Reliability and accuracy of fine-cut computed tomography scans to determine the status of anterior interbody fusions with metallic cages. Spine J. 2008 Nov-Dec;8(6):998-1002. doi: 10.1016/j.spinee.2007.12.004. Epub 2008 Feb 14. PMID 18280214